CLINICAL TRIAL: NCT00604006
Title: SCREEN-HFI (SCReening Evaluation of the Evolution of New Heart Failure Intervention Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: National Heart Foundation, Australia (Other)
Responsible Party: Principal Investigator, Prof Henry Krum, Prof Henry Krum, Monash University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CP-02/07
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure
Keywords: Prevention of heart failure in individuals at high risk
MeSH Terms: conditions — Heart Failure | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: Spironolactone
- Group B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — 25 mg tablets (placed in capsules for blinding) once daily.
  Arms: Group A
Drug: Placebo — Placebo (lactose in capsules for blinding) once daily
  Arms: Group B

SUMMARY:
Individuals who were a part of the investigators Screen-HF study (NCT00400257) whose BNP level are in the top quintile will be offered participation in this study. Participants will be randomised to receive either spironolactone or placebo for three years. Participants will then be monitored for indications of heart failure. It is anticipated that the medication will reduce the development of heart failure in this group.

ELIGIBILITY:
Inclusion Criteria:

1. Was recruited to SCREEN-HF
2. Has provided informed consent

Exclusion Criteria:

1. Uncorrected hyperkalaemia
2. eGFR < 30 ml/min

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Spironolactone in preventing heart failure | 1 year and 3 year
Cost effectiveness of Spironolactone prevention | 3 years

SECONDARY OUTCOMES:
Development of evidence of LV dysfunction, either systolic or diastolic, on echocardiography and/or symptomatic heart failure | 1 year and 3 year
Change in 6 minute walk test between the two groups | 1 year and 3 years
Change in quality of life between the two groups | 1 year and 3 year
Change in left ventricular remodelling parameters | 1 year and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS FRACP PhD, Principal Investigator — Monash University / Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Campbell DJ, Coller JM, Gong FF, McGrady M, Boffa U, Shiel L, Liew D, Stewart S, Owen AJ, Krum H, Reid CM, Prior DL. Kidney age - chronological age difference (KCD) score provides an age-adapted measure of kidney function. BMC Nephrol. 2021 Apr 26;22(1):152. doi: 10.1186/s12882-021-02324-y. PMID 33902478
- [Derived] Gong FF, Jelinek MV, Castro JM, Coller JM, McGrady M, Boffa U, Shiel L, Liew D, Wolfe R, Stewart S, Owen AJ, Krum H, Reid CM, Prior DL, Campbell DJ. Risk factors for incident heart failure with preserved or reduced ejection fraction, and valvular heart failure, in a community-based cohort. Open Heart. 2018 Jul 23;5(2):e000782. doi: 10.1136/openhrt-2018-000782. eCollection 2018. PMID 30057766